CLINICAL TRIAL: NCT02823093
Title: Aortic Calcification and Vitamin K Antagonists
Acronym: AVKAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0025
Record Dates: First submitted 2016-04-25; First posted 2016-07-06 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Vascular Calcification
Keywords: vascular calcification; aortic calcification; vitamin K antagonist; fluindione; warfarin; matrix gla protein
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A tube of blood on EDTA tubes of 6 ml will be taken at the elbow to the Clinical Research Center and then frozen at -80 ° . At the end of the study the tubes of all patients will be routed to VetAgro Sup Lyon in dry ice.
  DNA will be extracted from EDTA tubes . It will be stored frozen in the laboratory until analysis of polymorphisms of interest, by PCR technique .
  The promoter and the coding sequence of VKORC1 will be amplified by PCR and sequenced to detect the possible presence of SNPs
Oversight: Data Monitoring Committee: No

SUMMARY:
The vitamin K antagonists (VKA) are necessary drugs of prevention and treatment of thrombo-embolic disease. The AVKAL study assesses the impact of VKA treatment on the aortic calcifications development. This is a biomedical research without health product, transversal and monocentric study which compares the aortic calcifications levels of two populations : one treated by VKA and the other which has never been treated by VKA.

DETAILED DESCRIPTION:
The vitamin K antagonists exercise their anticoagulant effect by preventing the vitamin K dependant gamma-carboxylation of coagulation II, VII, IX and X factors which forms the final step of their activation.

They inhibit the vitamin K epoxide reductase VKORC1 enzyme, which is responsible of the vitamin K epoxide recycling in vitamin K hydroquinone (its reduced form). The carboxylation also can be inhibited by the Matrix Gla protein (MGP), inhibitor factor of vascular calcifications.

Warfarin (the most used VKA at the word level) is employed on animal for produce vascular calcifications by inhibiting the MGP activation.

Epidemiologic data indicate that warfarin could increase the calcifications of cardiac valves and coronary arteries. However, these studies were not interested in abdominal aorta's calcifications which are considered like an important marker of cardiovascular risk and did not concern the fluindione which is the most used VKA in France. Even if a class effect seems logical, the investigators can't dismiss the local effects, different to warfarin. In these studies, the calcifications assessment were rarely quantitative and the MGP levels were not measured. The vascular calcifications constitute a potential adverse effect of VKA which could limit their benefit in certain populations.

In this work there is an assumption that the aortic calcifications levels are upper in patients receiving VKA than in patients who are not receiving VKA and the aortic calcifications increase is owed to the non-activation of MGP.

The main objective is to assess if the taking of VKA is associated with the aortic calcifications development in patients receiving VKA.

Investigators will compare 2 populations: one group treated by VKA treatment for at least 6 months and one focus group which have never been treated by VKA treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients having a abdominal scanner without injection planned at CHU Amiens
* group treated by VKA: VKA treatment for at least 6 months
* group not treated by VKA: no antecedent of AVK treatment

Exclusion Criteria:

* abdominal scanner contre indication
* progressive cancer
* scanner planned by emergency department
* patient having had acute cardiovascular accident in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One group treated by VKA treatment for at least 6 months and one focus droup which have never been treated by VKA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Calcifications scores | at inclusion
  Agatston's method

SECONDARY OUTCOMES:
Plasmatic concentrations in dp-ucMGP | 12 months
  The first measure of MGP is actually a measure of the dephosphorylated MGP [ dpMGP ] performed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Cedric RENARD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Background] Price PA, Urist MR, Otawara Y. Matrix Gla protein, a new gamma-carboxyglutamic acid-containing protein which is associated with the organic matrix of bone. Biochem Biophys Res Commun. 1983 Dec 28;117(3):765-71. doi: 10.1016/0006-291x(83)91663-7. PMID 6607731
- [Background] Schurgers LJ, Aebert H, Vermeer C, Bultmann B, Janzen J. Oral anticoagulant treatment: friend or foe in cardiovascular disease? Blood. 2004 Nov 15;104(10):3231-2. doi: 10.1182/blood-2004-04-1277. Epub 2004 Jul 20. PMID 15265793
- [Background] Price PA, Faus SA, Williamson MK. Warfarin causes rapid calcification of the elastic lamellae in rat arteries and heart valves. Arterioscler Thromb Vasc Biol. 1998 Sep;18(9):1400-7. doi: 10.1161/01.atv.18.9.1400. PMID 9743228
- [Background] Schurgers LJ, Cranenburg EC, Vermeer C. Matrix Gla-protein: the calcification inhibitor in need of vitamin K. Thromb Haemost. 2008 Oct;100(4):593-603. PMID 18841280